CLINICAL TRIAL: NCT05257382
Title: A Randomized Controlled Study Evaluating the Added Value of an Hybrid Room Equipped With a Cone Beam CT (CBCT) to Electromagnetic Navigation Bronchoscopy (ENB) for the Diagnosis of Pulmonary Nodule.
Brief Title: Added Value of Cone Beam CT Guidance to Electromagnetic Navigation Bronchoscopy for the Diagnosis of Pulmonary Nodule.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Benjamin Bondue, Chest physician - MD PhD, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P2019/617
Record Dates: First submitted 2022-02-08; First posted 2022-02-25 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Lung Cancer; Pulmonary Disease
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endoscopy suite (Active Comparator): In this arm, ENB procedure will be performed in a classical endoscopy suite equipped by a fluoroscopy.
  Interventions: Procedure: ENB followed by trans-bronchial biopsy and trans-bronchial cryobiopsy
- CBCT suite (Experimental): In this arm, ENB procedure will be performed in a n hybrid room equipped by a cone beam CT (CBCT). This will allow to perform a real time visualisation of the lesion, enhanced fluoroscopy and to use the CrossCountry technique if required.
  Interventions: Procedure: ENB followed by trans-bronchial biopsy and trans-bronchial cryobiopsy

INTERVENTIONS:
Procedure: ENB followed by trans-bronchial biopsy and trans-bronchial cryobiopsy — After having performed the ENB procedure to reach the identified lung lesion, biopsies will be performed (six forceps trans-bronchial biopsies and one trans-bronchial lung cryobiopsy)

SUMMARY:
A monocentric prospective and randomized trial aiming to compare the diagnostic yield and safety of electromagnetical-guided bronchoscopy (ENB) procedures coupled to trans-bronchial lung cryobiopsies for the diagnosis of pulmonary nodule when performed either in a "standard" bronchoscopy suite or in a hybrid room with CBCT guidance and the use of the CrossCountry technique as required.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary nodule of maximum 30mm of largest diameter
* Nodules can be either solid or subsolid (including GGO) without evidence of loco-regional or distant metastasis that could be biopsied, and no evidence for an infectious underlying disease.
* A multidisciplinary discussion is performed for each case before considering its inclusion in the study in order to validate the indication of ENB-guided biopsy. Of note, any other endoscopic or trans-thoracic procedure should be tried before considering ENB if it could achieve the diagnosis according to the investigator's judgment.

Exclusion Criteria:

* Patient eligible for a direct surgical resection of the nodule
* Other exclusion criteria are a higher risk of bleeding (platelets count lower than 80,000/mm³, a systolic pulmonary arterial pressure (sPAP) higher than 45 mmHg at transthoracic ultrasonography, prothrombin time international normalized ratio - INR >1.5, activated partial thromboplastin time - APTT >35, uninterrupted anti-coagulant/anti-aggregant therapy), and the presence of any contraindication to general anesthesia as determined by the principal investigator (significant cardiac comorbidities, hypercapnia, severe hypoxia...).

No strict limits for inclusion were applied regarding diffusing capacity for carbon monoxide (DLCO), forced vital capacity (FVC), and forced expiratory volume in 1 second (FEV1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | Through study completion, an average of 1 year
  The primary outcome will be the comparison of the diagnostic yield obtained when ENB procedures will be performed on either the "classical " endoscopic suite or in the CBCT suite

SECONDARY OUTCOMES:
Rate of pneumothorax | up to 1 month after the procedure
  On the basis of control chest Xray performs after the endoscopic intervention. The need of chest drainage will also be recorded.
Rate of bleeding | up to 1 month after the procedure
  Bleeding will be scored as follows: score 0, when no bleeding occurs; score 1, when bleeding stops within five minutes either spontaneously or by inflation of a Fogarty balloon; score 2, when bleeding is prolonged more than five minutes or needs cold saline instillation; and score 3, when bleeding requires embolization, selective bronchial intubation, transfusion, admission in the intensive care unit, results in prolonged hospital stay, or patient's death.
Duration of the interventions | Up to one day after the procedure
  The total duration of the bronchoscope intervention will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bondue, PhD, Principal Investigator — Erasme University Hospital
Locations (1):
- Hopital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
When published, the datasets used and/or analysed during the study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the publication of the results
Access Criteria: The datasets used and/or analysed during the study will be available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Bondue B, Taton O, Tannouri F, Van de Velde N, Remmelink M, Leduc D. High diagnostic yield of electromagnetic navigation bronchoscopy performed under cone beam CT guidance: results of a randomized Belgian monocentric study. BMC Pulm Med. 2023 May 27;23(1):185. doi: 10.1186/s12890-023-02492-7. PMID 37245012